CLINICAL TRIAL: NCT04487366
Title: Comparison of Single and Double Operator Techniques in Ultrasound-guided Peripheral Nerve Block Learning Curve for Anesthesia Residency Training on a Gelatin-based Phantom Model: a Prospective Randomized Controlled Study
Brief Title: Single and Double Operator Techniques in Ultrasound-guided Peripheral Nerve Block Learning Curve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, ismail aytaç, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: E1/20-804
Record Dates: First submitted 2020-07-17; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Single-handed Ultrasound-guided Regional Anaesthesia Grip; Single-operator Ultrasound-guided Peripheric Nerve Block; Anesthesiology Training; Jedi Grip
Keywords: Jedi Grip; single-operator ultrasound-guided regional anaesthesia grip; Single-handed ultrasound-guided regional anaesthesia; 'On lock' grip; Anesthesiology training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Double Operator Ultrasound-Guided Regional Anesthesia (Active Comparator): resident control block needle and ultrasound probe and asistant operator inject the solution. resident reach the target area created in the phantom model using a block needle with ultrasound guidance
  Interventions: Other: reaching targeted area on the phantom model
- Jedi Grip (Active Comparator): resident control block needle, ultrasound probe and syringe independently with jedi grip; reach the target area created in the phantom model using a block needle with ultrasound guidance; inject and aspirate the solution.
  Interventions: Other: reaching targeted area on the phantom model
- On-lock grip (Active Comparator): resident control block needle, ultrasound probe and syringe independently with on-lock grip; reach the target area created in the phantom model using a block needle with ultrasound guidance; inject the solution.
  Interventions: Other: reaching targeted area on the phantom model
- Bedforth alternative grip (Active Comparator): resident control block needle, ultrasound probe and syringe independently with bedforth's alternative grip; reach the target area created in the phantom model using a block needle with ultrasound guidance; inject the solution.
  Interventions: Other: reaching targeted area on the phantom model

INTERVENTIONS:
Other: reaching targeted area on the phantom model — resident reach the targeted area on the phantom model using ultrasoun guidance and independently or with asistance inject the solution

SUMMARY:
Aim of this study is to compare learning curves of single(1- Jedi grip: Pappin and Christie/ 2- Bedforth/ 3- on lock: Gupta and Berrill) and double operator ultrasound-guided peripheric nerve block techniques on a home-made gelatin-based phantom model.

DETAILED DESCRIPTION:
Ultrasound-guided peripheral blocks are conventionaly performed by double operators. One operator controls both the ultrasound probe and peripheric block needle. Another assistant operator aspirate or injects local anesthetic. In this technique operator do not sense resistance in the syringe. Also this technique requires a well-done communication and coordination between operators.

In order to eliminate disadvantages of this technique several single-operator grip techniques of the needle and syringe have been described(1- Jedi grip: Pappin and Christie/ 2- Bedforth/ 3- on lock: Gupta and Berrill). Single operator techniques allow the provider to perform independently.

Aim of this study is to compare learning curves of single and double operator ultrasound-guided peripheric nerve block techniques on a home-made gelatin-based phantom model.

ELIGIBILITY:
Inclusion Criteria:

- To be a junior resident of anesthesiology(< 2 years )

Exclusion Criteria:

* Refusal of resident

Ages: 24 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-15 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Time to correct grip1 | during implementation of procedure on phantom model(first session)
  Time(sec) from start command to correct grip of the probe, needle and syringe for each technique
image quality1 | during implementation of procedure on phantom model(first session)
  provided image quality by resident for each technique which is assessed by investigator by four point Liker Scale( 1- much worse 2- worse 3- better 4- much better)
number of attempts1 | during implementation of procedure on phantom model(first session)
  number of attempts until correct needling to target area
needling time 1 | during implementation of procedure on phantom model(first session)
  time to reach target area with block needle
success of injection1 | during implementation of procedure on phantom model(first session)
  successful if injected water flows from hose of model/ unsuccessful if solution do not flow
Time to correct grip2 | during implementation of procedure on phantom model(second session)
  Time(sec) from start command to correct grip of the probe, needle and syringe for each technique
Time to correct grip3 | during implementation of procedure on phantom model(third session)
  Time(sec) from start command to correct grip of the probe, needle and syringe for each technique
image quality2 | during implementation of procedure on phantom model(second session)
  provided image quality by resident for each technique which is assessed by investigator by four point Liker Scale( 1- much worse 2- worse 3- better 4- much better)
image quality3 | during implementation of procedure on phantom model(third session)
  provided image quality by resident for each technique which is assessed by investigator by four point Liker Scale( 1- much worse 2- worse 3- better 4- much better)
number of attempts2 | during implementation of procedure on phantom model(second session)
  number of attempts until correct needling to target area
number of attempts3 | during implementation of procedure on phantom model(third session)
  number of attempts until correct needling to target area
needling time 2 | during implementation of procedure on phantom model(second session)
  time to reach target area with block needle
needling time 3 | during implementation of procedure on phantom model(third session)
  time to reach target area with block needle
success of injection2 | during implementation of procedure on phantom model(second session)
  successful if injected water flows from hose of model/ unsuccessful if solution do not flow
success of injection3 | during implementation of procedure on phantom model(third session)
  successful if injected water flows from hose of model/ unsuccessful if solution do not flow

SECONDARY OUTCOMES:
NASA-TLX (NASA Task Load Index) | during implementation of procedure on phantom model(third session)
  Resident assessment of each techniques for Mental Demand ,Physical Demand, Temporal Demand, Performance, Effort and Frustration
Assesment of education | during education of techniques
  Residents assesment of pre-procedural education with a questtionarie. "Education was sufficient enough to safely perform peripheral block":
  1. I absolutely agree
  2. I approve
  3. I am indecisive
  4. I do not approve
  5. Absolutely Disagree

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Aytac, Principal Investigator — Ankara City Hospital Anesthesiology Department
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pappin D, Christie I. The Jedi Grip: a novel technique for administering local anaesthetic in ultrasound-guided regional anaesthesia. Anaesthesia. 2011 Sep;66(9):845. doi: 10.1111/j.1365-2044.2011.06845.x. No abstract available. PMID 21831086
- [Background] Gupta P, Berrill A. 'On lock' - a further single-operator ultrasound-guided regional anaesthesia grip. Anaesthesia. 2017 Oct;72(10):1289. doi: 10.1111/anae.14050. No abstract available. PMID 28891057
- [Background] Bedforth N, Townsley P, Maybin J, Eisenberg E. Single-handed ultrasound-guided regional anaesthesia. Anaesthesia. 2011 Sep;66(9):846. doi: 10.1111/j.1365-2044.2011.06864.x. No abstract available. PMID 21831088
- [Background] Miyake S. Factors influencing mental workload indexes. J UOEH. 1997 Dec 1;19(4):313-25. doi: 10.7888/juoeh.19.313. PMID 9431583
- [Derived] Guven Aytac B, Unal S, Aytac I. A randomized, controlled simulation study comparing single and double operator ultrasound-guided regional nerve block techniques using a gelatine-based home-made phantom. Medicine (Baltimore). 2022 Sep 2;101(35):e30368. doi: 10.1097/MD.0000000000030370. PMID 36107586